CLINICAL TRIAL: NCT00039208
Title: Time Finding Study of Chronomodulated Irinotecan, 5 Fluorouracil, Leucovorin and Oxaliplatin as First or Second Chemotherapy Line Against Metastatic Colorectal Cancer
Brief Title: Combination Chemotherapy in Treating Patients With Colorectal Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: European Organisation for Research and Treatment of Cancer - EORTC (Network)
Responsible Party: Sponsor
Allocation: Randomized | Purpose: Treatment
Other Study IDs: EORTC-05011; EORTC-05011
Record Dates: First submitted 2002-06-06; First posted 2003-01-27 (Estimated); Last update posted 2012-07-13 (Estimated); Status verified 2012-07

CONDITIONS: Colorectal Cancer
Keywords: stage III colon cancer; stage IV colon cancer; stage III rectal cancer; stage IV rectal cancer; recurrent colon cancer; recurrent rectal cancer
MeSH Terms: conditions — Colorectal Neoplasms; Colonic Neoplasms; Rectal Neoplasms | interventions — Fluorouracil; Irinotecan; Leucovorin; Oxaliplatin

INTERVENTIONS:
Drug: fluorouracil
Drug: irinotecan hydrochloride
Drug: leucovorin calcium
Drug: oxaliplatin

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die. Giving drugs at the time of day that allows for the best drug response may allow the doctor to give higher doses of chemotherapy drugs and kill more tumor cells.

PURPOSE: Randomized phase II trial to determine the best time to give irinotecan combined with fluorouracil, leucovorin, and oxaliplatin in treating patients who have colorectal cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the role of peak delivery time on the tolerability of irinotecan when administered with chronomodulated fluorouracil, leucovorin calcium, and oxaliplatin as first- or second-line therapy in patients with locoregional or metastatic colorectal cancer.
* Determine the antitumor activity of this regimen.

OUTLINE: This is a randomized, multicenter study. Patients are stratified according to participating center, WHO performance status (0-1 vs 2), and line of treatment (first vs second). Patients are randomized to receive irinotecan at 1 of 6 different times of the day.

Patients receive irinotecan IV over 6 hours on day 1 and fluorouracil IV and leucovorin calcium IV over 11 hours followed by oxaliplatin IV over 11 hours on days 2-5. Courses repeat every 21 days in the absence of disease progression or unacceptable toxicity.

Patients are followed every 4 weeks until disease progression and then every 8 weeks thereafter.

PROJECTED ACCRUAL: A maximum of 186 patients (31 per irinotecan administration time) will be accrued for this study within 2 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed colorectal cancer
* Unresectable metastatic or locoregional disease
* At least 1 measurable lesion outside a previously irradiated area or an area treated with physical devices (e.g., cryotherapy, laser, or thermoablation)
* No prior enrollment in EORTC-05963
* No symptomatic brain metastases

PATIENT CHARACTERISTICS:

Age:

* Over 18

Performance status:

* WHO 0-2

Life expectancy:

* Not specified

Hematopoietic:

* Neutrophil count greater than 2,000/mm^3
* Platelet count at least 90,000/mm^3

Hepatic:

* Bilirubin no greater than 2 times upper limit of normal (ULN)

Renal:

* Creatinine no greater than 1.5 times ULN
* No uncontrolled hypercalcemia

Cardiovascular:

* No overt cardiac disease

Pulmonary:

* No severe respiratory illness

Other:

* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception
* Male patients must use effective barrier contraception during and for up to 6 months after study
* No baseline diarrhea greater than grade I (must have less than 4 stools per 24 hours)
* No prior grade III or IV toxicity related to irinotecan
* No sensory or motor neuropathy with functional impairment
* No prior hypersensitivity to any study drug
* No other primary tumor except basal cell skin cancer or carcinoma in situ of the cervix
* No uncontrolled infectious or chronic disease
* No psychological, familial, sociological, or geographical condition that would preclude study

PRIOR CONCURRENT THERAPY:

Biologic therapy:

* No concurrent prophylactic growth factor therapy

Chemotherapy:

* At least 1 month since prior chemotherapy
* No prior irinotecan, fluorouracil, leucovorin calcium, and oxaliplatin as combination therapy
* Other prior therapy containing irinotecan and/or oxaliplatin allowed
* No more than 1 prior chemotherapy regimen for metastatic or locoregional disease
* Adjuvant chemotherapy considered first-line therapy if tumor relapsed within 6 months of completion of therapy

Endocrine therapy:

* No concurrent corticosteroids except for emergencies

Radiotherapy:

* See Disease Characteristics
* Palliative radiotherapy for bone lesion allowed except for disease progression

Surgery:

* See Disease Characteristics

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 2002-02; Primary Completion 2005-08 (Actual)

PRIMARY OUTCOMES:
Peak delivery time for CPT11 tolerability over the first 3 courses of treatment in patients who started therapy

SECONDARY OUTCOMES:
Peak delivery time for CPT11 tolerability over the first 3 courses of treatment in patients who started therapy, excluding those who stopped prior to course 3 for reasons other than toxicity
Peak delivery time for CPT11 activity over the first 3 courses
Peak delivery time for CPT11 tolerability and efficacy over the first 6 courses
Severe toxic events assessed by CTC v2.0 after each course of chemotherapy
Progression-free survival
Overall survival

CONTACTS AND LOCATIONS:
Overall Officials: Carlo Garufi, MD, Study Chair — Istituti Fisioterapici Ospitalieri - Roma
Locations (20):
- Belgium (5):
  - Centre Hospitalier Notre Dame - Reine Fabiola, Charleroi
  - Clinique Saint-Joseph, Liège
  - CHU Liege - Domaine Universitaire du Sart Tilman, Liège
  - Clinique Sainte Elisabeth, Namur
  - Centre Hospitalier Peltzer-La Tourelle, Verviers
- France (6):
  - Centre Jean Perrin, Clermont-Ferrand
  - Centre de Lutte Contre le Cancer Georges-Francois Leclerc, Dijon
  - Centre Hospital Regional Universitaire de Limoges, Limoges
  - Hopital Saint-Louis, Paris
  - Centre Rene Huguenin, Saint-Cloud
  - Hopital Paul Brousse, Villejuif
- Italy (8):
  - Azienda Sanitaria di Bolzano, Bolzano
  - Universita G.D'Annunzio Di Chieti, Chieti
  - Ospedale San Carlo Borromeo, Milano (Milan)
  - Azienda Ospedale S. Luigi at University of Torino, Orbassano, (Torino)
  - Fondazione Salvatore Maugeri, Pavia
  - Ospedale Oncologico Regionale, Rionero in Vulture
  - Istituto Regina Elena, Rome
  - Istituto Clinico Beato Matteo, Vigevano
- Hospital Fernando Fonseca, Amadora, Portugal

REFERENCES:
- [Result] Garufi C, Focan C, Tumolo S, et al.: Time finding study of chronomodulated irinotecan (I), fluorouracil (F), leucovorin (L) and oxaliplatin (O) (chronoIFLO) against metastatic colorectal cancer: results from randomized EORTC 05011 trial. [Abstract] J Clin Oncol 25 (Suppl 18): A-2566, 2007.